CLINICAL TRIAL: NCT01629901
Title: The Effect of Vestibular Stimulation on Cerebral Blood Flow
Brief Title: Caloric Stimulation on Cerebral Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Scion NeuroStim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00035775
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2015-06

CONDITIONS: Healthy Volunteer
Keywords: Healthy volunteer
MeSH Terms: interventions — Neoplasm Staging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ThermoNeuroModulation (TNM) Device — Non-invasive neurostimulator used for up to 20 minutes in a session.

SUMMARY:
This is a prospective, non-randomized study designed to generate preliminary data to assess the effect of a new portable non-invasive caloric stimulator on EEG waveform and cerebral blood flow on normal healthy volunteers.

DETAILED DESCRIPTION:
Study activities include monitoring with bilateral transcranial Doppler (TCD), EEG and continuous EKG monitoring at 30 second intervals for 5 minutes. This is followed by placement of the caloric stimulator investigational device for 20 minutes. An additional 20 minutes of TCD and EEG monitoring will also be recorded. This will end study participation.

ELIGIBILITY:
Inclusion Criteria:

* no history of neurological disease

Exclusion Criteria:

* persons under the age of 18
* pregnant or nursing women
* history of neurological disease
* history of psychiatric disease
* congenital heart defect, known cardiac shunt
* inner ear or pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Changes in cerebral blood flow | 20 minutes
  Changes in cerebral blood flow will be quantified through the use of bilateral transcranial Doppler (TCD). The baseline TCD of three vessels will be compared with measurements taken at 30 second intervals for 5 minutes after caloric stimulation.

SECONDARY OUTCOMES:
Alterations in EEG readings | 40 minutes
  EEG readings occurring between baseline, active CVS induction, and post-CVS induction periods will be assessed to identify and characterize alterations in the readings.
Alterations in regional cerebral brain flow (rCBF) | 40 minutes
  A standard noninvasive near infrared spectroscopy system will be used to look for any alterations in rCBF induced by CVS treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Laskowitz, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States